CLINICAL TRIAL: NCT04463043
Title: The Effectiveness of an App-based (selfBACK) Versus a Web-based (e-Help) Self-management Intervention or Usual Care in People With Low Back and/or Neck Pain on a Waiting List for Hospital-based Outpatient Rehabilitation: a Three Arm Randomised Controlled Trial
Brief Title: An App-based Versus a Web-based Self-management Intervention or Usual Care in People With Low Back and/or Neck Pain on a Waiting List for Hospital-based Outpatient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 64084
Record Dates: First submitted 2020-06-18; First posted 2020-07-09 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Back Pain; Neck Pain
Keywords: self-management; rehabilitation; mHealth; eHealth
MeSH Terms: conditions — Back Pain; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is a single-blinded trial. Participants and health personnel at the clinic will not be blinded to group allocation, whereas researchers performing the analysis and the interpretation of the results will be blinded to group allocation. Once the study is completed, the data will be extracted from the database in anonymized form for statistical analyses, i.e. all personal information that may identify specific participants or group allocation will be removed and the intervention and control groups will be randomly labelled as A, B and C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SelfBACK app (Experimental): The selfBACK app in addition to usual care
  Interventions: Device: SelfBACK app; Other: Usual care
- e-Help webpage (Active Comparator): The e-Help webpage in addition to usual care
  Interventions: Other: e-Help webpage; Other: Usual care
- Usual care (Active Comparator): Usual care only
  Interventions: Other: Usual care

INTERVENTIONS:
Device: SelfBACK app — The selfBACK is an evidence-based and data-driven decision support system (DSS) to support self-management of low back and neck pain delivered via a smartphone app. The selfBACK app provides individually tailored self-management plans to participants on a weekly basis by matching the participant's health information with targeted educational messages, physical activity advices and exercise recommendations via the DSS.
  Arms: SelfBACK app
Other: e-Help webpage — The e-Help is an evidence-based web-based resource to support self-management of low back and neck pain. The e-Help webpage provides evidence-based self-management content equivalent to the selfBACK including educational messages, physical activity and exercise recommendations. Instructions on how to compose exercise programs will be given to participants, however no tailored self-management support will be offered in this solution.
  Arms: e-Help webpage
Other: Usual care — Usual care refers to seeking care or receiving treatments or help as usual.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an individually tailored self-management intervention, the selfBACK app, in improving health status in patients on a waiting list for outpatient rehabilitation due to low back and/or neck pain compared to a non-tailored web-based self-management solution (e-Help) and usual care only.

DETAILED DESCRIPTION:
Patients on waiting list for treatment at the multidisciplinary outpatient clinic for back, neck and shoulder rehabilitation, St. Olavs Hospital, Trondheim University Hospital, Norway, due to low back and/or neck pain are the target group for this study. The average waiting time for receiving treatment is 8-10 weeks. The use of digital solutions can be a beneficial approach to support self-management during the waiting period. Therefore, the effectiveness of these tools in this patients group needs to be evaluated.

A total of 279 participants will be recruited and randomly allocated to one of the three groups: 1) the selfBACK app in addition to usual care; 2) the e-Help webpage in addition to usual care; and 3) usual care only. Participants who receive either the selfBACK app and the e-Help webpage will be allowed to seek care, treatment or help elsewhere as usual.

Self-reported outcome measures will be collected through web-based questionnaires at three follow-up time points: 1) 6 weeks; 2) 3 months (primary endpoint); and 3) 6 months. In addition, participants receiving the selfBACK app will be asked a set of weekly tailoring questions to individualize self-management plans. Objective registry based data linked to social security number in Norway will be used to investigate health care consumption and sickness absence at 1 year (and up to 5 years).

ELIGIBILITY:
Inclusion Criteria:

* On waiting list for treatment at the multidisciplinary outpatient clinic for back, neck and shoulder rehabilitation, St. Olavs Hospital, Trondheim University Hospital, Norway due to low back pain and/or neck pain
* Own and use a smartphone with internet access to download the mobile application
* Able to provide informed consent

Exclusion Criteria:

* Less than 4 weeks waiting time until scheduled appointment at clinic (i.e., patients prioritized for urgent treatment/examination)
* Unable to take part in exercise/physical activity, e.g. non-ambulatory patients, use of walking aids, unable to get up and down the floor independently
* Unable to speak and/or read Norwegian
* Unable to complete the baseline questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal Health Questionnaire (MSK-HQ) | Change from baseline to 3 months
  The MSK-HQ is used to measure musculoskeletal health status. The MSK-HQ contains 14 items scored from 0 to 4. The final score ranges from 0 to 56 (sum of all items), with higher scores indicating better musculoskeletal health status.

SECONDARY OUTCOMES:
Pain-related disability for low back pain | Change from baseline to 3 months
  Pain-related disability is measured by the Roland Morris Disability Questionnaire (RMDQ) ranging from 0 to 24. Higher scores indicate higher pain-related disability.
Pain-related disability for neck pain | Change from baseline to 3 months
  Pain-related disability is measured by the Neck Disability Index (NDI) ranging from 0 to 50. Higher scores indicate higher pain-related disability.
Average pain intensity | Change from baseline to 3 months
  The average pain intensity within the past week is measured by a 11-point numerical rating scale (NRS) ranging from 0='no pain' to 10='worst pain imaginable'.
Worst pain intensity | Change from baseline to 3 months
  The worst pain intensity within the past week is measured by a 11-point numerical rating scale (NRS) ranging from 0='no pain' to 10='worst pain imaginable'.
Health related quality of life | Change from baseline to 3 months
  The EuroQoL 5-dimension (EQ-5D) questionnaire is used to assess health-related quality of life. 5 items scored 0 - 5 plus visual analogue scale scored 0- 100.
Pain self-efficacy | Change from baseline to 3 months
  The Pain Self-Efficacy Questionnaire (PSEQ) is used to assess participants' level of confidence in carrying out specific activities despite their pain. 10 items scored 0 - 6.
Illness perception | Change from baseline to 3 months
  The Brief Illness Perception Questionnaire (BIPQ) is used to evaluate participants' illness perception. 8 items scored 0 - 10.

OTHER OUTCOMES:
Fear avoidance belief | Change from baseline to 3 months
  The Fear-Avoidance Belief Questionnaire (FABQ) - physical activity subscale is used to measure participant's beliefs about how physical activity affect their low back and/or neck pain. 5 items scored 0 - 6
Stress symptoms | Change from baseline to 3 months
  The Perceived Stress Scale (PSS) is used to evaluate stress levels. 10 items scored 0 - 4.
Depressive symptoms | Change from baseline to 3 months
  The Patient Health Questionnaire-2 (PHQ-2) is used to evaluate patients' depressive symptoms. 2 items scored 0 - 3.
Functional change | Change from baseline to 3 months
  The Patient Specific Functional Scale (PSFS) is used to evaluate changes in participant's ability to perform up to two self-selected activities regarded as important by them. Ability levels scored 0 - 10.
Self-reported physical activity | Change from baseline to 3 months
  The modernised Saltin-Grimby Physical Activity Level Scale is used to evaluate self-reported leisure time physical activity. 1 item (4 options).
Self-reported sleep | Change from baseline to 3 months
  Sleep problems are assessed by four self-report items which provide information needed to diagnose insomnia according to the DSM-V criteria. 4 items scored 0 - 2.
Work ability | Change from baseline to 3 months
  Work ability index (WAI) is used to assess work ability. 1-item rated on an 11-point numeric rating scale (0='completely unable to work' to 10='work ability at its best').
Satisfaction with intervention | 3 months
  Patient Acceptable Symptom State (PASS) is used to determine if patients consider themselves well and, as such, are satisfied with the treatment. 1 item (yes/no)
Perceived effect | 3 months
  Patient's Global Perceived Effect is used to investigate participants' perception of effect from the intervention they received. 1 item scored -5 to 5
Health care consumption | 1 year
  Objective registry based data linked to social security number in Norway are used to investigate health care consumption.
Sickness absence | 1 year
  Objective registry based data linked to social security number in Norway are used to investigate sickness absence.

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Tverrfaglig poliklinikk rygg/nakke/skulder, St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available, including data dictionaries. Data available to share include individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 5 years after end of trial and ending 30 years after end of trial.
Access Criteria: Investigators whose proposed use of the data has been approved by the national ethics committee. Proposals should be directed to the principal investigator. To gain access, data requestors will need to sign a data access agreement. Information regarding submitting proposals and accessing data may be found at (Link will be provided after completing the trial).

REFERENCES:
- [Background] Marcuzzi A, Bach K, Nordstoga AL, Bertheussen GF, Ashikhmin I, Boldermo NO, Kvarner EN, Nilsen TIL, Marchand GH, Ose SO, Aasdahl L, Kaspersen SL, Bardal EM, Borke JB, Mork PJ, Gismervik S. Individually tailored self-management app-based intervention (selfBACK) versus a self-management web-based intervention (e-Help) or usual care in people with low back and neck pain referred to secondary care: protocol for a multiarm randomised clinical trial. BMJ Open. 2021 Sep 13;11(9):e047921. doi: 10.1136/bmjopen-2020-047921. PMID 34518253
- [Derived] Marcuzzi A, Klevanger NE, Aasdahl L, Gismervik S, Bach K, Mork PJ, Nordstoga AL. An Artificial Intelligence-Based App for Self-Management of Low Back and Neck Pain in Specialist Care: Process Evaluation From a Randomized Clinical Trial. JMIR Hum Factors. 2024 Jul 9;11:e55716. doi: 10.2196/55716. PMID 38980710
- [Derived] Marcuzzi A, Nordstoga AL, Bach K, Aasdahl L, Nilsen TIL, Bardal EM, Boldermo NO, Falkener Bertheussen G, Marchand GH, Gismervik S, Mork PJ. Effect of an Artificial Intelligence-Based Self-Management App on Musculoskeletal Health in Patients With Neck and/or Low Back Pain Referred to Specialist Care: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2320400. doi: 10.1001/jamanetworkopen.2023.20400. PMID 37368401